CLINICAL TRIAL: NCT00656266
Title: A Prospective Randomized Trial of Prednisone and Tacrolimus Versus Prednisone, Tacrolimus and Mycophenolate Mofetil in Pediatric Liver Transplantation
Brief Title: Trial of Calcineurin Inhibitor-Sparing Immunosuppression Regimen in Pediatric Liver Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient funding
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, John Goss, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-15138
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: End-stage Liver Disease; Renal Insufficiency; Renal Failure
Keywords: renal insufficiency or failure; liver transplantation
MeSH Terms: conditions — End Stage Liver Disease; Renal Insufficiency | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- tacrolimus & corticosteroids (Placebo Comparator): Standard post-transplant immunosuppression medications: tacrolimus and corticosteroids
  Interventions: Other: placebo medication
- low-dose tacrolimus + steroids + MMF (Experimental): Comparison arm: low-dose tacrolimus + steroids + MMF
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — immunosuppresion medication called mycophenolate mofetil, also known as MMF or CellCept
  Other Names: CellCept; MMF
  Arms: low-dose tacrolimus + steroids + MMF
Other: placebo medication — medication that looks like mycophenolate mofetil
  Other Names: placebo pill
  Arms: tacrolimus & corticosteroids

SUMMARY:
The objective of this study is to compare the effects of two liver transplant immunosuppression regimens on renal function. Patients receiving the standard combination of prednisone and high-dose tacrolimus, a drug with known nephrotoxicity (Arm A) will be compared to patients receiving prednisone, low-dose tacrolimus and mycophenolate mofetil (MMF) (Arm B). MMF is an immunosuppression agent that has no associated nephrotoxicity. The primary end point of the study will be renal function as measured by glomerular filtration rate (GFR). Thirty pediatric liver transplant recipients will be randomized to these two arms in a 1:1 ratio (i.e. 15 patients in each group). Secondary end points will measure patient and graft outcome and incidence of immunosuppression-related complications, including: neurotoxicity, diabetes mellitus, growth retardation, vomiting, diarrhea, gastrointestinal hemorrhage, thrombocytopenia, anemia, leukopenia, acute or chronic liver graft rejection, posttransplant lymphoproliferative disease (PTLD), viral infections, fungal infections and bacterial infections.

DETAILED DESCRIPTION:
The objective of this study is to compare the effects of two liver transplant immunosuppression regimens on renal function. Patients receiving the standard combination of prednisone and high-dose tacrolimus, a drug with known nephrotoxicity (Arm A) will be compared to patients receiving prednisone, low-dose tacrolimus and mycophenolate mofetil (MMF) (Arm B). MMF is an immunosuppression agent that has no associated nephrotoxicity. The primary end point of the study will be renal function as measured by glomerular filtration rate (GFR). Thirty pediatric liver transplant recipients will be randomized to these two arms in a 1:1 ratio (i.e. 15 patients in each group). Secondary end points will measure patient and graft outcome and incidence of immunosuppression-related complications, including: neurotoxicity, diabetes mellitus, growth retardation, vomiting, diarrhea, gastrointestinal hemorrhage, thrombocytopenia, anemia, leukopenia, acute or chronic liver graft rejection, posttransplant lymphoproliferative disease (PTLD), viral infections, fungal infections and bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* End-stage liver disease or acute fulminant hepatic failure recalcitrant to conventional medical or surgical therapy.
* Listed as candidate for pediatric liver transplantation listed with United Network for Organ Sharing (UNOS).
* Patients must be 18 years of age or younger.

Exclusion Criteria:

* History of autoimmune disease or primary sclerosing cholangitis.
* History of end-stage renal disease, dialysis treatment or acute renal failure (not including hepatorenal syndrome).
* Patients with pretransplant renal insufficiency as determined by a glomerular filtration rate (GFR) of <80 mL/min/1.73m2 (see below).
* Patients with renal agenesis or hypoplasia, polycystic kidney disease, or hydroureter seen on pretransplant renal ultrasound.
* Patients with malignancy or previous malignancy.
* Patients with active bacterial, viral, or fungal infections.
* Patients with a pretransplant diagnosis of diabetes mellitus.
* Patients with history of previous transplant or multi-organ recipients.
* Patients with serological evidence of HIV, HBSAg or HCV.
* Patients with hereditary syndrome that causes genetic deficiency of hypoxanthine-guanine phosphoribosyl-transferase (HGPRT) such as Lesch-Nyhan or Kelley-Seegmiller syndrome.
* Patients with history of phenylketonuria.
* Females that are pregnant or breastfeeding.
* Sexually active females who are not: a) post-menopausal, or b) surgically sterile, and c) using an acceptable method of contraception (oral contraceptive, implanted devices, injection, and barrier devices are acceptable; condoms used alone are not acceptable).
* Patients with alcohol abuse, substance abuse or smoking within the previous 6 months.
* Patients or caretakers of patients with psychogenic factors that preclude therapeutic compliance.
* Inability to reach participating hospital within 2 hours of notification.
* Any conditions or any circumstance that makes it unsafe to undergo a liver transplant.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2004-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
change in glomerular filtration rate (GFR) two years after liver transplantation as calculated by the Schwartz formula | two years
  change in glomerular filtration rate (GFR) two years after liver transplantation as calculated by the Schwartz formula

CONTACTS AND LOCATIONS:
Overall Officials: John Goss, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States